CLINICAL TRIAL: NCT03393676
Title: Preoperative Chronic Pain Increases the Risk of Early Postoperative Cognitive Dysfunction in Elderly Patients Undergoing Hip Joint Replacement Surgery: a Prospective Observational Cohort Study
Brief Title: Preoperative Pain and POCD in Elderly Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Xiaorong Huai, Dr., RenJi Hospital
Other Study IDs: PPOCD20161201
Record Dates: First submitted 2017-12-26; First posted 2018-01-08 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Postoperative Cognitive Dysfunction
Keywords: Postoperative Cognitive Dysfunction; elderly patients; Preoperative Pain
MeSH Terms: conditions — Postoperative Cognitive Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to investigate whether preoperative pain is the risk factor of POCD in elder patients.

DETAILED DESCRIPTION:
Postoperative cognitive dysfunction (POCD) occurs mainly in aged patients. The mechanism of POCD is not clear yet and no effective therapy method. In the present study, we conducted a single-center observational prospective cohort trial in elder patients who undergoing hip joint replacement surgery with general anesthesia to test our hypothesis that preoperative chronic pain is one of the risk factors of POCD after major joint replacement surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Elder than 65 years old
2. Speak Chinese Mandarin
3. Those who will undergo major low limb surgery like hemiarthroplasty or total hip arthroplasty with general anesthesia.
4. Signed the inform consent
5. American Society of Anesthesiologists classification I to II

Exclusion Criteria:

1. Existing cerebral disease, or have a history of neurological and psychiatric disease including Alzheimer Disease, stroke, epilepsy and psychosis
2. Existing cognitive impairment as evidenced by Mini-Mental State Examination scores below 24
3. Severe hearing or visual impairment
4. Unwillingness to comply with the protocol or procedures
5. Cannot communicate with Chinese Mandarin
6. Serious pulmonary, heart , liver or renal insufficiency patients
7. Had anesthesia or surgery within the past 30 days

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly patients underwent elective low limb surgery(hemiarthroplasty or total hip arthroplasty); Chronic pain duration >3 months.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-01-10 (Actual); Primary Completion 2020-03-31 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
POCD incidence 7 days (or before leaving hospital) after surgery | 7 days (or before leaving hospital)
  POCD incidence 7 days (or before leaving hospital) after surgery

SECONDARY OUTCOMES:
POCD incidence 2 months after surgery | 2 months after surgery
  POCD incidence 2 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Weifeng Yu, MD, Study Chair — Anesthesiology Department Renji Hospital, Shanghai
Locations (2):
- China (2):
  - Reni Hospital, Shanghai Jiao Tong University, School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Ren ji Hospital, Shanghai, Shanghai Municipality

REFERENCES:
- [Derived] Huai X, Jiao Y, Gu X, Zhu H, Chen L, Fan Y, Yu W, Su D, Xie H. Preoperative Chronic Pain as a Risk Factor for Early Postoperative Cognitive Dysfunction in Elderly Patients Undergoing Hip Joint Replacement Surgery: A Prospective Observational Cohort Study. Front Neurosci. 2021 Dec 17;15:747362. doi: 10.3389/fnins.2021.747362. eCollection 2021. PMID 34975369